CLINICAL TRIAL: NCT02472756
Title: Relapsed/Refractory Follicular Lymphoma - Rituximab Therapy in Combination With Chemotherapy
Brief Title: A Study of Rituximab in Combination With Chemotherapy in Relapsed/Refractory Follicular Lymphoma
Acronym: REFLECT 2
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21872
Record Dates: First submitted 2015-05-28; First posted 2015-06-16 (Estimated); Results first posted 2016-08-12 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Drug Therapy; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Follicular Lymphoma Participants: Previously treated adult participants with relapsed/refractory FL will receive rituximab in combination with chemotherapy regimen. All treatments prescribed during the observation period will be at the treating physician's discretion. Participants will be followed up for safety and efficacy evaluation in accordance with routine practice, up to 30 months.
  Interventions: Drug: Chemotherapy; Drug: Rituximab

INTERVENTIONS:
Drug: Chemotherapy — The choice of the chemotherapy regimen will be established on a per center basis, according to the standard in use in the country and in the center. Protocol does not specify any particular chemotherapy regimen.
Drug: Rituximab — The choice of the rituximab regimen will be established on a per center basis, according to the standard in use in the country and in the center. Protocol does not specify any particular chemotherapy regimen.
  Other Names: MabThera

SUMMARY:
This is a Phase 4, open, prospective, non-interventional, multicenter trial for previously treated adult participants with relapsed/refractory follicular lymphoma (FL). Eligible participants with FL will receive 6-8 infusions of induction standard regimen of rituximab plus chemotherapy. Participants with complete or partial remission at end of induction will be assigned to maintenance therapy with rituximab once every 3 months for a maximum of 2 years or until relapse. The choice of the treatment regimen will be established on a per center basis, according to the standard in use in the country and in the center, and each center will use the same regimen through the study. Participants will be followed up for safety and efficacy evaluation in accordance with routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with FL and had already received one or more treatments

Exclusion Criteria:

* Participants who are not eligible for rituximab treatment according to summary of product characteristics (SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously treated adult participants with relapsed/refractory FL
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2008-09-19 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2014-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Serbia (6):
  - Institute of Hematology, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - Institute For Oncology Sremska Kamenica; Internal Medicine Department, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
  - Clinic of Haematology Cc Nis, Niš
  - Clinical Center Vojvodine; Clinic for Hematology, Novi Sad

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All treatments prescribed during the observation period were at the treating physician's discretion and should have been prescribed according to package labeling, within approved indication and local approval status of respective drugs.
Groups:
- Follicular Lymphoma Participants: Previously treated adult participants with relapsed/refractory follicular lymphoma received induction treatment with rituximab in combination with chemotherapy regimen for approximately 6 months followed by maintenance therapy with rituximab for a maximum of 2 years. All treatments prescribed during the observation period were at the treating physician's discretion. Participants were followed up for safety and efficacy evaluation in accordance with routine practice, up to 30 months.
Period: Induction (Approximately 6 Months)
Arm/Group | Follicular Lymphoma Participants
Started | 41
Treated | 40
Completed | 39
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Enrolled But Not Treated | 1
Period: Maintenance (Approximately 2 Years)
Arm/Group | Follicular Lymphoma Participants
Started | 20 (Out of 39 participants who completed induction period, 19 did not continue in maintenance period.)
Completed | 10
Not Completed | 10
Not completed — Lack of Drug | 7
Not completed — Progression Disease | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all treated participants.
Arm/Group | Follicular Lymphoma Participants
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 55 [40 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response
Description: Lymphoma response was assessed using Cheson criteria. Objective response was defined as having either complete remission (CR) or partial remission (PR). Criteria for CR (target lesions): Nodes returned to normal (if greatest transverse diameter [GTD] greater than [>] 15 millimeters [mm] before therapy, GTD now less than or equal to [≤] 15 mm; if GTD 11-15 mm and short axis [SA] >10 mm before therapy, SA now ≤10 mm) and all (non-nodal) target lesions completely resolved. Criteria for CR (non-target lesions): All non-target lymph nodes returned to normal size, all extra-nodal lesions have completely resolved, liver and spleen have returned to normal size (if enlarged at baseline). Criteria for PR: Sum of the product of the diameters (SPD) of target lesions decreased at least 50 percent (%) from baseline and spleen and liver nodules regressed by 50% in SPD or single lesion in GTD.
Time Frame: Baseline until disease progression or death, whichever occurred first (up to approximately 6 months)
Population: Intent-to treat (ITT) population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Follicular Lymphoma Participants
Number analyzed (Participants) | 39
percentage of participants | 92.3

2. Primary Outcome: Percentage of Participants With Complete Remission (CR)
Description: Lymphoma response was assessed using Cheson criteria. Criteria for CR (target lesions): Nodes returned to normal (if GTD >15 mm before therapy, GTD now ≤15 mm; if GTD 11-15 mm and SA >10 mm before therapy, SA now ≤ 10 mm) and all (non-nodal) target lesions completely resolved. Criteria for CR (non-target lesions): All non-target lymph nodes returned to normal size, all extra-nodal lesions have completely resolved, liver and spleen have returned to normal size (if enlarged at baseline).
Time Frame: Baseline until disease progression or death, whichever occurred first (up to approximately 6 months)
Population: ITT population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Follicular Lymphoma Participants
Number analyzed (Participants) | 39
percentage of participants | 56.4

3. Primary Outcome: Percentage of Participants Who Were Alive at Year 2
Time Frame: Year 2
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Follicular Lymphoma Participants
Number analyzed (Participants) | 40
percentage of participants | 85

ADVERSE EVENTS:
Time Frame: Up to 30 months
Arm/Group | Follicular Lymphoma Participants
Serious Adverse Events (participants affected / at risk) | 8/41
Other Adverse Events (participants affected / at risk) | 3/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Follicular Lymphoma Participants (N=41)
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Leukemias acute myeloid (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Hypogammaglobulinaemia (Immune system disorders) | 1
Tracheitis (Respiratory, thoracic and mediastinal disorders) | 1
Hepatitis B (Infections and infestations) | 1
Death (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Follicular Lymphoma Participants (N=41)
Neutropenia (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.